CLINICAL TRIAL: NCT07007338
Title: Calcium Isotope Ratios to Assess Calcium Bone Balance in Dialysis Children Receiving Cinacalcet - The Cin-Ca Study
Brief Title: Calcium Isotope Ratios to Assess Calcium Bone Balance in Dialysis Children Receiving Cinacalcet
Acronym: Cin-ca
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_1148
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Children Over 3 Undergoing Dialysis With Secondary Hyperparathyroidism
Keywords: CKD-MBD; children; secondary hyperparathyroism; Cinacalcet; dialysis
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood : 1 to 3 tubes per visit / 4 visits Urines : 1 tube per visit / 4 visits
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children above 3 years of age on maintenance dialysis who begin treatment with cinacalcet: Children above 3 years of age on maintenance dialysis (hemodialysis, hemodiafiltration, peritoneal dialysis) who begin treatment with cinacalcet because of secondary hyperparathyroism
  Interventions: Biological: Supplementary blood samples and urines samples

INTERVENTIONS:
Biological: Supplementary blood samples and urines samples — Supplementary blood and urines samples realised during routine visits

SUMMARY:
Managing bone and mineral disorders associated with chronic kidney disease (CKD-MBD) in children is a complex task. Controlling parathyroid hormone (PTH) levels involves adjusting calcium intake, managing hyperphosphatemia, intensive dialysis, and considering specific therapies like active vitamin D analogues and cinacalcet.

Cinacalcet, authorized in Europe since 2017 for children over 3 undergoing dialysis with secondary hyperparathyroidism (SHPT), has shown efficacy in reducing PTH levels. The 2019 guidelines call for its use with caution particularly to avoid hypocalcemia, in children with severe hyperparathyroidism despite optimized conventional treatments.

In adults, cinacalcet has been found to reduce serum PTH, calcium, and phosphate levels, decrease the risk of vascular calcification, and have a positive effect on bone formation. This suggests that cinacalcet may slow the progression of cardiovascular calcifications.

Additionally, Professor Shroff has introduced a non-invasive method for assessing bone calcium status by analyzing stable calcium isotope ratios in blood. This method would allow to determine whether a treatment such as cinacalcet has a positive influence on bone calcium balance, a key element in the management of CKD-MBD.

ELIGIBILITY:
Inclusion Criteria:

* Children from 3 to 17 years of age
* On maintenance dialysis : hemodialysis, hemodiafiltration, peritoneal dialysis
* Patient who begin treatment with cinacalcet based on the 2019 European guidelines and at the discretion of the treating physician
* With normal QTc interval on electrocardiogram
* With total serum calcium >2.40 mmol/L
* With heamoglobin > 8g/dl
* Non - opposition from parents/legal guardians

Exclusion Criteria:

* Children < 12 kg
* Persons deprived of their liberty by a judicial or administrative decision
* Persons under psychiatric care
* Persons admitted to a health or social institution for purposes other than research
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
* Persons participating in other interventional research with an exclusion period still in progress at pre-inclusion
* Patients who received cinacalcet with 3 months prior inclusion

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will involve children above 3 years of age on maintenance dialysis (hemodialysis, hemodiafiltration, peritoneal dialysis) who begin treatment with cinacalcet.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
value of isotope ratios of calcium (44/42 Ca) in blood | Baseline / 3 months treatment
  value of 44/42 Ca ratio in patients at baseline and, three months after cinacalcet treatment

CONTACTS AND LOCATIONS:
Overall Officials: BACCHETTA Justine, MD, Principal Investigator — Hospices Civils de Lyon
Locations (7):
- France (7):
  - Service de Pédiatrie CHU de Bordeaux, Bordeaux
  - Hôpital Femme Mère Enfant, Bron
  - Service de pédiatrie multidisciplinaire CHU de Montpellier, Montpellier
  - Unité de néphrologie pédiatrique, Hôpital Archet 2, CHU de Nice, Nice
  - Service de Néphrologie pédiatrique Hôpital Necker Enfants Malades, Paris
  - Service de Néphrologie - Transplantation - Hémodialyse pédiatrique Hôpital Robert Debré, Paris
  - Service de pédiatrie 1 CHU Hautepierre, Strasbourg

IPD SHARING:
Plan to Share IPD: No